CLINICAL TRIAL: NCT01389453
Title: Umbilical Cord Mesenchyma Stem Cell Transplantation in Patients With Cerebral Hemorrhage and Cerebral Infarction
Brief Title: The Clinical Trial Research of Stem Cell Transplantation Treats Cerebral
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: There were not enough number of patients recruited till DEC 31th in 2012.
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2011-04-17 stroke
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2011-10

CONDITIONS: Stroke
Keywords: umbilical cord mesenchyma stem cell transplantation
MeSH Terms: conditions — Stroke | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stem cell transplatation (Active Comparator): All experimental group patients accept a treatment course stem cell transplantation, including one time stem cell transplantation through intravenous injection way at the 10-21th day of cerebral hemorrhage, and the 7-14th day of cerebral infarction incidence; the second time transplantation through lumbar puncture way at the 7th day after the First time transplantation.
  Interventions: Procedure: stem cell transplantation
- control (No Intervention): The control group gives injection through intravenous and lumbar puncture ways separately in the corresponding time, but the transplantation matter is physiological saline not the stem cell.

INTERVENTIONS:
Procedure: stem cell transplantation — Patients accept a treatment course stem cell transplantation, including one time stem cell transplantation through intravenous injection way at the 10-21th day of cerebral hemorrhage, and the 7-14th day of cerebral infarction incidence; the second time transplantation through lumbar puncture way at the 7th day after the First time transplantation.
  Other Names: umbilical cord mesenchyma stem cell transplantation
  Arms: stem cell transplatation

SUMMARY:
All experimental group patients of 100 patients accept a treatment course stem cell transplantation, including one time stem cell transplantation through intravenous injection way at the 10-21th day of cerebral hemorrhage, and the 7-14th day of cerebral infarction incidence; the second time transplantation through lumbar puncture way at the 7th day after the First time transplantation. The control group gives injection through intravenous and lumbar puncture ways separately in the corresponding time, but the transplantation matter is physiological saline not the stem cell.

DETAILED DESCRIPTION:
The control group of 20 patients accept injection through intravenous and lumbar puncture ways separately in the corresponding time, but the transplantation matter is physiological saline not the stem cell.

ELIGIBILITY:
Inclusion Criteria:

1. All tested patients with cerebral infarction, cerebral hemorrhage must tally with the diagnosis standard which in 1995 the Chinese fourth session of brain blood vessel of academic conference formulated, and after the head CT, MRI confirmation. All patients should be taken bad completely within for 24 hours.
2. patient's age and gender: 40-65years，the gender is not limit;
3. the hemorrhage, block region：One side basis festival area, one side brain stem;
4. the patient must catch the apoplexy at the first time and the accidence causes the obvious clinical symptoms.

Exclusion Criteria:

1. Progressive apoplexy;
2. other internal organs strict illness sickness, like serious heart disease, diabetes, liver, kidney vigorous sickness and so on;
3. the patient with tumor in every system on there body;
4. Having the primary or the sequential epilepsy medical history, within one year had the epileptic paroxysm;
5. can not accept MRI inspection, for some metal implant in there body(such as inner support in heart or brain blood vessel).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
NIHSS and FIM | before the transplant and after the transplant 1, 2 and 3 months
  All patients should receive the American State-run Health Research institute apoplexy meter (NIHSS)evaluation, the Fugl-Meyer evaluation, the function independence evaluation (FIM) separately before the transplant and after the transplant 1, 2 and 3 months , and the grading has the distinct improvement;

SECONDARY OUTCOMES:
Motor evoked potential and sensation evoked potential inspection | before the transplant and after the transplant 0, 1, 3, 6 and 12 months
  All patients should be receive Motor evoked potential and sensation evoked potential inspection separately before the transplant and after the transplant 0, 1, 3, 6 and 12 months, and the function of movement and sensation get obvious improvement;
MRI+ DWI+ enhancement scanning | before the transplant and after the transplant 0, 1, 3, 6 and 12 months
  All patients should be receive cranial MRI+ DWI+ enhancement scanning separately before the transplant and after the transplant 0, 1, 3, 6 and 12 months, and the result tells us that there is obvious blood vessel proliferation on the surrounding of damaged region;

CONTACTS AND LOCATIONS:
Overall Officials: An Yihua, doctor, Study Director — Chinese People's Armed Police Force
Locations (1):
- Yihua An, Beijing, Beijing Municipality, China